CLINICAL TRIAL: NCT05152433
Title: E-BRAiN - Evidence-Based Robot-Assistant in Neurorehabilitation
Brief Title: Evidence-Based Robot-Assistant in Neurorehabilitation
Acronym: E-BRAiN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: BDH-Klinik Greifswald (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202101E-BRAiN; CIV-21-01-035629 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2021-11-07; First posted 2021-12-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Paresis; Neglect, Hemispatial
MeSH Terms: conditions — Stroke; Paresis; Perceptual Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Length of period: 2 weeks
  Interventions: Behavioral: Conventional therapy
- Therapy assisted by a humanoid robot (E-BRAiN) (Experimental): Length of period: 2 weeks Fixed dose: 10 therapy sessions with E-BRAiN
  Interventions: Device: E-BRAiN therapy

INTERVENTIONS:
Device: E-BRAiN therapy — The therapy system E-BRAiN is a purpose-built therapy system using a socially interactive humanoid robot and provides individualised therapy for arm rehabilitation based on the evidence-based therapies arm basis training, arm ability training, or mirror therapy for arm rehabilitation (paresis) or neurovisual training (neglect).
  Arms: Therapy assisted by a humanoid robot (E-BRAiN)
Behavioral: Conventional therapy — Conventional therapy specifies the neurorehabilitation therapy as applied as regular treatment.
  Arms: Conventional therapy

SUMMARY:
The purpose of this study is to investigate the efficacy, acceptability, and safety of the therapeutic system E-BRAiN for the treatment of stroke-related impairments.

DETAILED DESCRIPTION:
This randomized controlled trial, RCT with cross-over design sequentially allocates participants with stroke-related impairment to both a two week course of conventional rehabilitation therapy and a two week course of therapy using the therapy system E-BRAiN (purpose-built therapy system using a socially interactive humanoid robot); participants are randomly allocated to the sequences "conventional => robot" or "robot => conventional". Stroke survivors with one of the target syndromes, i.e. mild arm paresis, or moderate to severe arm paresis, or visuospatial neglect are invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Age at study entry ≥ 18 years
* Stroke (ischemic stroke, non-traumatic intracerebral haemorrhage, subarachnoidal haemorrhage)
* Incomplete arm paresis (Motricity Index, arm score >1 [Min] and < 100 [Max]) or
* Visuospatial neglect (clinical signs and NET subtest "star cancellation" score < 50)
* Candidate able to consent and provides informed consent or
* legal representative provides informed consent

Exclusion Criteria:

* Pregnant or breast feeding
* Obliged to live in an institution by law or public authority
* With case presentation arm paresis: another condition that causes arm paresis is present
* With case presentation visuospatial neglect: another condition that causes a relevant visual-perceptual deficit that cannot be compensated is present; exception: homonymous visual field deficits are not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change scores over two weeks for the standardised primary outcome measure | 2 weeks
  Change scores are difference scores for assessments taken two weeks apart. Changes scores are based on standardised outcome measures. Assessment scores for each measure (see below) are standardised using the known variance in stroke survivor populations for the respective measure.
  The following assessments will be used for standardised outcome measures:
  Nine-Hole-Peg-Test, NHPT (finger dexterity) and Box-and-Block Test, BBT (gross manual dexterity) (for participants with mild arm paresis); Fugl Meyer, Arm motor score, FM Arm (selective arm and hand movement capacity) (participants with moderate to severe arm paresis); Neglect-Test, NET (spatial visual attention) (participants with visual neglect).

SECONDARY OUTCOMES:
Drop-out rate | 2 weeks
  Drop-outs
Goal attainment | 2 weeks
  Goal attainment Scale (GAS)
Change scores over two weeks for "Motivation for therapy" | 2 weeks
  Change scores are difference scores for assessments taken two weeks apart with Visual Analogue Scales (VAS) for motivational factors (Min 0, Max 100)
Change scores over two weeks for "Emotional distress" | 2 weeks
  Change scores are difference scores for assessments taken two weeks apart with the Hospital Anxiety and Depression Scale (HADS)
Work alliance | 2 weeks
  Assessment of the perceived work alliance for the period of two weeks prior using the Work Alliance Inventory (WAI)
Adverse events | 2 weeks
  Adverse events documentation for the period of two weeks

OTHER OUTCOMES:
Type and frequency of neurorehabilitation therapy received | 2 weeks
  Therapy documentation for the period of two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Platz, Prof.Dr.med., Principal Investigator — Head, Neurorehabilitation Research Group
Locations (2):
- Germany (2):
  - Universitätsmedizin Greifswald, Greifswald
  - BDH-Klinik Greifswald, Greifswald

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Research web site — http://www.ebrain-science.de/en/home/